CLINICAL TRIAL: NCT02795117
Title: Comparative Safety and Efficacy of Two Treatments in the Treatment of Inflammatory Lesions of Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-15-013
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test product (Experimental)
  Interventions: Drug: Ivermectin
- Reference product (Active Comparator)
  Interventions: Drug: Ivermectin (reference)
- Placebo product (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin
  Arms: Test product
Drug: Ivermectin (reference)
  Arms: Reference product
Drug: Placebo
  Arms: Placebo product

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Perrigo's product to an FDA approved product for the treatment of inflammatory lesions rosacea

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an Institutional Review Board (IRB) approved written informed consent for this study.
2. Must be at least 18 years of age
3. Must have a definite clinical diagnosis of moderate to severe facial papulopustular rosacea
4. Subjects must be willing and able to understand and comply with the requirements of the study and apply the medication as instructed.
5. Subjects must be in general good health and free from any clinically significant disease, other than rosacea, that might interfere with the study evaluations.
6. Females of childbearing potential (excluding women who are surgically sterilized (verified tubal ligation or bilateral oophorectomy or hysterectomy) or post- menopausal for at least 2 years), in addition to having a negative urine pregnancy test at Visit 1/Day 1 (Baseline), must be willing to use an acceptable form of birth control during the study.

Exclusion Criteria:

1. Subjects, who are pregnant, breastfeeding, or planning a pregnancy within the period of their study participation.
2. Current or past ocular rosacea.
3. Presence of any other facial skin condition that might interfere with rosacea diagnosis and/or assessment.
4. History of hypersensitivity or allergy to the study medication and/or any ingredient in the study medication.
5. Use of radiation therapy and/or anti-neoplastic agents within 90 days prior to Visit 1/Day 1 (Baseline).
6. Current use of anticoagulation therapy and use throughout the study.
7. Use of medicated make-up (including anti-aging make-up) throughout the study
8. Use during the study of 1) systemic steroids, 2) topical retinoids to the face 3) antibiotics known to impact rosacea 4) immunosuppressive agents, or immunomodulators).
9. Facial use of 1) topical steroids, 2) topical anti-inflammatory agents, 3) topical antimycotics, 4) any topical rosacea treatments or 4) topical antibiotics.
10. Use of medicated cleansers on the face (throughout the study.
11. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements
12. Use of topical astringents or abrasives, medicated topical preparations (prescription and OTC products) within 2 days prior to Visit 1 and throughout the study.
13. Use of antipruritics (including antihistamines), spa treatments or chlorine exposure (swimming etc.) within 24 hours of all study visits.
14. Participation in any clinical study involving an investigational product, agent or device that might influence the intended effects or mask the side effects of study medication in the 1 month (30 days) prior Visit 1/Day 1 (Baseline) or throughout the study.
15. Previous enrollment in this study or current enrollment in this study at another participating site.
16. Use of tanning booths, sun lamps (excessive UV radiation e.g., phototherapy, daily extended exposure or occupational exposure to the sun), sunbathing or excessive exposure to the sun 1 week prior to baseline and throughout the study.
17. Subjects who in the opinion of the investigator, are unlikely to be able to follow the restrictions of the protocol and complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: Ivermectin cream
- Reference Product: Ivermectin (reference) cream
- Placebo: Placebo cream
Period: Overall Study
Arm/Group | Test Product | Reference Product | Placebo
Started | 193 | 193 | 100
Completed | 175 | 166 | 88
Not Completed | 18 | 27 | 12

BASELINE CHARACTERISTICS:
Groups:
- Test Product: Ivermectin Cream, 1% (Perrigo)
- Reference Product: Ivermectin Cream, 1% (reference)
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Placebo | Total
Number analyzed (Participants) | 193 | 193 | 100 | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.65) | 51.3 (13.61) | 51.2 (14.25) | 51.5 (13.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 140 | 67 | 348
  Male | 52 | 53 | 33 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 37 | 19 | 94
  Not Hispanic or Latino | 155 | 156 | 81 | 392
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 0 | 0 | 2 | 2
  White | 188 | 189 | 97 | 474
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in the Inflammatory (Papules and Pustules) Lesion Count
Time Frame: Day 1 to Day 84
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of lesion reduction
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 156 | 147 | 75
percentage of lesion reduction | 65.47 (30.222) | 67.89 (30.244) | 55.51 (32.660)
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — provides 85% power of success; ANOVA — No p-value was calculated for bioequivalence, only a T/R ratio and 90% confidence interval; equivalence ratio = 96.4, 90% CI 2-sided [91.0 to 105.4]

2. Secondary Outcome: Subjects With Clinical Success on the Investigator Global Assessment
Description: Clinical success is defined as a score of clear or almost clear
Time Frame: Day 1 to Day 84
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Test Product | Reference Product | Placebo
Number analyzed (Participants) | 156 | 147 | 75
Participants | 71 | 79 | 26
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Equivalence — provides 85% power of success; Wald's method; Equivalence difference = -6.48, 90% CI 2-sided [-18.31 to 1.85]

ADVERSE EVENTS:
Time Frame: Day 1 to day 84
Arm/Group | Test Product | Reference Product | Placebo
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/193 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/193 | 0/193 | 0/100
Other Adverse Events (participants affected / at risk) | 0/193 | 0/193 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT02795117/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT02795117/SAP_001.pdf